CLINICAL TRIAL: NCT04439123
Title: MATCH Treatment Subprotocol Y: AZD5363 in Patients With Tumors With AKT Mutations
Brief Title: Testing AZD5363 as a Potential Targeted Treatment in Cancers With AKT Genetic Changes (MATCH-Subprotocol Y)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-02980; NCI-2020-02980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Y (Other: ECOG-ACRIN Cancer Research Group); EAY131-Y (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (capivasertib) (Experimental): Patients receive capivasertib PO BID on days 1-4, 8-11, 15-18, and 22-25. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — Given PO
  Other Names: AZD 5363; AZD-5363; AZD5363; Truqap

SUMMARY:
This phase II MATCH treatment trial identifies the effects of AZD5363 in patients whose cancer has a genetic change called AKT mutation. AZD5363 may block AKT, which is a protein needed for cancer cell growth. Researchers hope to learn if AZD5363 will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive capivasertib (AZD5363) orally (PO) twice daily (BID) on days 1-4, 8-11, 15-18, and 22-25. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have an AKT mutation as determined via the MATCH Master Protocol
* Patients with hormone receptor positive, defined as estrogen receptor and/or progesterone receptor > 1% by immunohistochemistry, AND HER2 negative unresectable breast cancer, with no overexpression by immunohistochemistry (IHC) or amplification by in-situ hybridization, are allowed to continue fulvestrant or an aromatase inhibitor (anastrozole, letrozole, exemestane) with AZD5363 if patient just progressed on this anti-estrogen therapy. Gonadotrophin releasing hormone (GnRH) agonists (such as leuprolide or goserelin) are allowed. For instance, if the last treatment was letrozole plus goserelin, the patient is allowed to continue the letrozole plus goserelin with AZD5363

  * NOTE: Selective estrogen receptor modulators (SERMs), such as tamoxifen or toremifene, are not allowed, given concerns about CYPD26 and CYP3A4 metabolism, respectively
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with diabetes or risk for hyperglycemia are eligible. Patients with diabetes mellitus may enter the study unless any of the following exclusion criteria are fulfilled:

  * Baseline fasting glucose value of > 8.9 mmol/L or 160 mg/dL (fasting is defined as no calorific intake for at least 8 hours)
  * Insulin required for routine diabetic management and control
  * More than two oral hypoglycemic medications required for routine diabetic management and control

Exclusion Criteria:

* Patients must not have known hypersensitivity to AZD5363 or compounds of similar chemical or biologic composition
* Patients with known KRAS, NRAS, HRAS, or BRAF mutations are not eligible for this protocol, as these mutations may lead to limited response due to resistance
* Patients may not have received treatment with another inhibitor of PI3K, AKT or mTOR in the neoadjuvant, adjuvant or metastatic setting with the exception of FDA approved rapalogs. Patients with metastatic cancer, who received PI3K/AKT/mTOR inhibitors on short preoperative window trials (treatment for 4 weeks or less) will be eligible if the treatment was over 6 months prior to registration
* Patients may not have received strong inhibitors or potent inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Kalinsky, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] McCourt CK, Gross J, Kalinsky K, Guan P, McShane LM, Wang V, O'Dwyer PJ, Lahey MT, Maican C, Bu X, Patton D, Harris LN. Comprehensive Molecular and Genomic Analysis of NCI-MATCH Subprotocol Y: Capivasertib in Patients With an AKT1 E17K-Mutated Tumor. JCO Precis Oncol. 2025 Mar;9:e2400614. doi: 10.1200/PO-24-00614. Epub 2025 Mar 28. PMID 40153687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Y was activated on May 31, 2016. A total of 43 patients were assigned to this arm after screening, 42 from screening cohort and 1 from outside assay. Of the 43 patients, 35 patients were enrolled to arm Y between July 13, 2016 and August 10, 2017.
Pre-assignment Details: To be assigned to a specific MATCH subprotocol, patients needed to submit a tumor biopsy for molecular characterization and those with molecular variants addressed by treatments included in the trial entered corresponding MATCH subprotocol. For the subprotocol Y, patients had to have an AKT mutation.
Period: Overall Study
Arm/Group | Treatment (Capivasertib)
Started | 35 (All 35 patients enrolled were eligible and treated in the arm)
Completed | 0
Not Completed | 35
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Disease progression | 19
Not completed — Withdrawal by Subject | 2
Not completed — Still on treatment | 2

BASELINE CHARACTERISTICS:
Population: Patients who were eligible and received protocol treatment
Arm/Group | Treatment (Capivasertib)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 61 [32 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) among all eligible and treated patients. Best overall response was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. The 90% two-sided binomial exact confidence interval was calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Capivasertib)
Number analyzed (Participants) | 35
percentage of participants | 28.6 [15 to 46]

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Patients who were eligible and received protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Capivasertib)
Number analyzed (Participants) | 35
percentage of participants | 50 [35 to 71]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Patients who were eligible and received protocol treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Capivasertib)
Number analyzed (Participants) | 35
months | 5.5 [4.6 to 11.3]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All 35 cases that received protocol treatment were monitored for adverse events.
Arm/Group | Treatment (Capivasertib)
All-Cause Mortality (participants affected / at risk) | 23/35
Serious Adverse Events (participants affected / at risk) | 20/35
Other Adverse Events (participants affected / at risk) | 29/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Capivasertib) (N=35)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Capivasertib) (N=35)
Anemia (Blood and lymphatic system disorders) | 4
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 6
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 6
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 11
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04439123/Prot_001.pdf